CLINICAL TRIAL: NCT03249987
Title: Comparing the Usability of an Electronic Bladder Diary and a Paper Bladder Diary: a Two-way Crossover Study
Brief Title: Comparing the Usability of an Electronic Bladder Diary and a Paper Bladder Diary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STH19309
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2017-08

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic bladder diary (Other): Participants will be asked to complete the electronic diary for three days before crossing over to the paper diary. Patients will be asked to record the time and volume of voids, any incontinence or urgency episodes and sleep-wake times. Patients will be asked to complete a short questionnaire regarding their opinions
  Interventions: Other: bladder diary
- Paper bladder diary (Other): Participants will be asked to complete the paper diary for three days before crossing over to the electronic diary. Patients will be asked to record the time and volume of voids, any incontinence or urgency episodes and sleep-wake times. Patients will be asked to complete a short questionnaire regarding their opinions
  Interventions: Other: bladder diary

INTERVENTIONS:
Other: bladder diary — electronic diary to be completed for 3 days before crossover onto paper diary for 3 days

SUMMARY:
This piece of research is a single centre, two-way cross over, prospective study to compare the outcomes and experience of patients completing a paper bladder diary and an electronic version. This project aims to examine whether an electronic bladder diary can improve data quality compared to a paper bladder diary. Participants will attend an introduction appointment within the Urology Department at Royal Hallamshire Hospital. The participant will complete the bladder diaries at home and will then complete a questionnaire at the Royal Hallamshire Hospital.

Patients who are being sent an appointment for urodynamics (standard or video) will be also sent a recruitment letter and participant information sheet (PIS), to inform them of the study. One week later a member of the study team will phone the patient, to see if they are interested in participating in the study and assess the eligibility criteria. If that patient is interested and they fulfil the inclusion/exclusion criteria they will be invited to attend an introduction appointment. This will be conducted 1-2 weeks prior to the urodynamic test, at which point study details will be discussed and written informed consent will be taken. The participant will be taught how to use the digital and paper versions of the bladder diaries

Participants will be asked to complete the electronic diary for three days and the paper diary for three days. Half of the participants will complete the digital diary first, the other half will complete the paper diary first, and this will be done by alternating consecutively. Patients will be asked to record the time and volume of voids, any incontinence or urgency episodes and sleep-wake times. On the day of their urodynamics appointment, patients should return with their electronic and paper diaries

DETAILED DESCRIPTION:
Micturition time-charts, frequency-volume charts and bladder diaries are inexpensive, non-invasive tools that allow the assessment of lower urinary tract symptoms (Konstantinidis et al. 2011); with a large proportion of women giving them low burden scores (Vella et al. 2012).

A micturition time chart records 'the times of micturitions, day and night, for at least 24 hours' (Abrams et al. 2002), whereas frequency-volume charts record 'the volumes voided as well as the time of each micturition, day and night, for at least 24 hours' (Abrams et al. 2002) and a bladder diary 'records the times of micturitions and voided volumes, incontinence episodes, pad usage and other information such as fluid intake, the degree of urgency and the degree of incontinence' (Abrams et al. 2002). However, the three terms are often used interchangeably in the literature, purely meaning documentation of void time, volume and +/- urgency.

Frequency-volume charts are used to record patients' symptoms before and after therapeutic interventions and in bladder training, to assess the success of the treatment (Abrams and Klevmark, 1996).

NICE (2013) states that men with bothersome lower urinary tract symptoms should complete a urinary frequency-volume chart as part of their initial assessment. They provide information on: daytime frequency, nocturia, 24-hour frequency, 24-hour production, polyuria, nocturnal urine volume, nocturnal polyuria and maximum voided volume (Abrams et al. 2002). Frequency-volume charts can help to distinguish between nocturnal polyuria and detrusor overactivity by assessing the volume of urine voided (NICE, 2013).

Frequency-volume charts provide an insight in a patient's voiding patterns in their own environment and during their usual daily activities (Konstantinidis et al. 2011). A high test-retest reliability been shown for frequency-volume charts (Jimenez-Cidre et al. 2015; Yap et al. 2007), demonstrating their dependability.

The use of a frequency-volume chart can reduce recall error (Locker et al. 2001), as when retrospectively assessed >50% of patients overestimated daytime frequency in comparison to their frequency-volume chart (Stav et al. 2009).

Electronic diaries have been trailed in other areas of healthcare, most with success. Electronic diaries used to monitor asthma symptoms (Jiang et al. 2009), pain (Stone et al. 2003), headaches (Allena et al. 2012), amongst others showed to have a higher compliance compared to paper diaries.

Stone et al. (2003) compared the completion of a paper and electronic pain diary. The paper diary was fitted with a hidden device to track the opening and closing of the binder, to help monitor completion. It was found that on 32% of study days the paper diary was not opened, yet the compliance for these days was >90%. This suggests there has been backfilling of data, questioning the reliability of the data. This is further confirmed by Gaertner et al. (2004) who demonstrated more retrospective fabrication of data in the paper diary.

Broderick (2008) suggested that the time taken for data analysis is significantly reduced when using an electronic diary compared to a paper diary. However, the time for software installation and training should be taken into consideration.

A pain monitoring study showed that electronic diaries had a higher rate of compliance and less back dating of information (Stone et al. 2003).

Despite a number of patients lacking experience in the use of computers, patient satisfaction was higher for the electronic diary in a number of studies (Gaertner et al. 2004; Broderick, 2008), with many saying it was easy to understand and to use (Allena et al. 2012)

This is a single centre, two-way cross over, prospective study to compare the outcomes and experience of patients completing a paper bladder diary and an electronic version.Participants will attend an introduction appointment within the Urology Department at Royal Hallamshire Hospital. The room will ensure privacy for the patient. The participant will complete the bladder diaries at home. The participant will complete the questionnaire at the Royal Hallamshire hospital, in private.Participants will be asked to complete the electronic diary for three days and the paper diary for three days. Half of the participants will complete the digital diary first, the other half will complete the paper diary first, and this will be done by alternating consecutively.

Patients will be asked to record the time and volume of voids, any incontinence or urgency episodes and sleep-wake times. Patients return one week later with their electronic and paper diaries. Patients will be asked to complete a short questionnaire regarding their opinions. Clinicians should analyse the data as usual. Introduction and follow-up appointments will try to be arranged around patients' hospital appointments to avoid additional visits. Patients will be provided with an ELAROS electronic bladder diary as the electronic diary.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years old
* Patients must speak, read and write English
* Willing to participate in the study and able to provide written informed consent

Exclusion Criteria:

• Patients with limited verbal and/or written communication problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
The comparability between diary types | 3 days
  Number of days with more than one entry

SECONDARY OUTCOMES:
The comparability of the data values obtained from the electronic bladder diary and the paper bladder diary for Mean daytime frequency of urination | 6 days
  average daytime frequency
Patient satisfaction and preference of the electronic bladder diary against the paper diary. | 6 days
  Whether a patient prefers using the electronic diary over the paper diary as measure by the patient preference questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Richard Inman, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Royal Hallamshire Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD